CLINICAL TRIAL: NCT01391754
Title: Effectiveness Trial for Project SafeCare for Child Neglect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency); Oklahoma Department of Health and Human Services (Unknown)
Responsible Party: Mark Chaffin, PhD - Principal Investigator, University of Oklahoma Health Sciences Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 5R01MH065667 (NIH)
Record Dates: First submitted 2011-06-29; First posted 2011-07-12 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Child Neglect
Keywords: child abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SafeCare with Coached Implementation (Experimental): Home-based services with the SafeCare model, implemented with in vivo provider coaching as quality control
  Interventions: Behavioral: SafeCare; Other: In vivo coached quality control
- SafeCare without Coaching (Experimental): Home-based services using the SafeCare model, implemented without in vivo coached implementation quality control
  Interventions: Behavioral: SafeCare; Other: Uncoached
- Services As Usual with Coaching (Experimental): Usual home based services, with in vivo coached implementation quality control
  Interventions: Other: In vivo coached quality control; Behavioral: Services As Usual
- Services As Usual Without Coaching (Active Comparator): Usual home based services without in vivo coached quality control
  Interventions: Behavioral: Services As Usual; Other: Uncoached

INTERVENTIONS:
Behavioral: SafeCare — Behavioral home based family preservation. Weekly visits X six months.
  Arms: SafeCare with Coached Implementation; SafeCare without Coaching
Other: In vivo coached quality control — Live observation of practice with expert coaching, feedback and fidelity monitoring
  Arms: SafeCare with Coached Implementation; Services As Usual with Coaching
Behavioral: Services As Usual — Home based services not using the SafeCare model
  Arms: Services As Usual Without Coaching; Services As Usual with Coaching
Other: Uncoached — No in vivo coached quality control or fidelity monitoring
  Arms: SafeCare without Coaching; Services As Usual Without Coaching

SUMMARY:
The study is a field trial comparing the SafeCare family preservation model to a comparable usual care model for parents in child welfare. The study also compares two levels of service quality control.

DETAILED DESCRIPTION:
The study is a cluster-randomized field trial of the SafeCare(SC) home-based family preservation model for families in the child welfare system. The trial is conducted in collaboration with the state child welfare agency and their contracted in-home service system. The service system is regionalized and provides in home services to families referred by child welfare. Regions of the state are assigned by the study to either the SC model or to services as usual. Provider teams, nested within regions, are assigned to either a monitored or unmonitored model implementation quality control condition. The aims of the project are to test client level child welfare reentry outcomes between SC and standard conditions, across the two implementation and quality control conditions.

ELIGIBILITY:
Inclusion Criteria:

* Parents in the child welfare system for neglect with or without physical abuse

Exclusion Criteria:

* Parents in the child welfare system for sexual abuse

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2175 (Actual)
Dates: Start 2003-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Child welfare system recidivism | Up to 2766 days
  Follow-up for recidivism reports to child welfare, captured from administrative data maintained by the state child welfare system

SECONDARY OUTCOMES:
Child Abuse Potential Inventory | Approximately 180 days and 365 days
  This is a questionnaire survey measuring parenting distress, parenting attitudes, and risk for committing child abuse
Family Resources Scale | Approximately 180 and 365 days
  This is a questionnaire survey measuring sufficiency of basic concrete resources in a family, such as adequate food, shelter, utilities, clothing, access to health care, etc.
Beck Depression Inventory | Approximately 180 and 365 days
  This is a questionnaire measuring symptoms of depression
Social Provisions Scale | Approximately 180 and 356 days
  This is a questionnaire measuring the degree of social support and quality of social relationships
Diagnostic Interview Schedule--Drug and Alcohol Disorders Module | Approximately 180 and 365 days
  This is a structured diagnostic psychiatric interview, adapted to questionnaire format, measuring symptoms of alcohol disorders and drug disorders, with associated DSM based diagnostic algorithms.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Chaffin, PhD, Principal Investigator — University of Oklahoma
Locations (3):
- United States (3):
  - Eastern Oklahoma Youth Services, McAlester, Oklahoma
  - NorthCare, Oklahoma City, Oklahoma
  - Family and Children's Services, Tulsa, Oklahoma

REFERENCES:
- [Result] Aarons GA, Sommerfeld DH, Hecht DB, Silovsky JF, Chaffin MJ. The impact of evidence-based practice implementation and fidelity monitoring on staff turnover: evidence for a protective effect. J Consult Clin Psychol. 2009 Apr;77(2):270-80. doi: 10.1037/a0013223. PMID 19309186
- [Result] Chaffin M, Bard D. Changes in parental depression symptoms during family preservation services. Child Abuse Negl. 2011 Jun;35(6):448-58. doi: 10.1016/j.chiabu.2011.02.005. Epub 2011 Jun 1. PMID 21632109
- [Result] Chaffin M, Bard D, Hecht D, Silovsky J. Change trajectories during home-based services with chronic child welfare cases. Child Maltreat. 2011 May;16(2):114-25. doi: 10.1177/1077559511402048. Epub 2011 Apr 13. PMID 21493617